CLINICAL TRIAL: NCT05339698
Title: 3D Evaluation to Quantify Regional Volume Change Between FRC and TLC
Acronym: MATH3D
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220330; 2021-A02798-33 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Diaphragmatic Dysfunction
Keywords: Neuromuscular; Diaphragm; Non invasive; 3D analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is first to validate an IC measurement using analysis of two 3D acquisitions, and to appreciate the inter-observer variability of this IC measurement between a trained technician of respiratory function analysis and a trained pulmonologist.

DETAILED DESCRIPTION:
3D visualization of the chest and abdomen surface in static condition is a simple and inexpensive solution to measure regional volume changes between two static respiratory volume positions. Five seconds of apnea is necessary for visualizing the thoraco-abdominal surface. If the two positions visualized correspond to the functional residual capacity (FRC) and the total lung capacity (TLC) the volume difference is inspiratory capacity (IC) which depends to the inspiratory muscles activation. This IC can be split in different thoraco-abdominal compartments and in supine position the abdominal contribution of this IC volume appreciates non-invasively diaphragmatic function. In addition asymmetry between right and left sides can appreciate unilateral diaphragmatic.

The aim of this study is first to validate an IC measurement using analysis of two 3D acquisitions, and to appreciate the inter-observer variability of this IC measurement between a trained technician of respiratory function analysis and a trained pulmonologist.

Accordingly, patients addressed for suspicion of diaphragmatic dysfunction, and able to maintain 5 sec of apnea in supine position will be proposed, by using the informed consent process, to participate to this study which consisted to beneficiate to a 3D trunk visualization at FRC and TLC during a spirometric IC measurement in supine position. Thoraco-abdominal volume difference between the two positions (FRC and TLC) will be calculated to obtain a 3D-IC volume. Then a Bland-Altman comparison will be done between the 3D-IC volumes measured and calculated by the two different observers (technician and pulmonologist), and the spirometric-IC volume considered as the reference. The Bland-Altman average discrepancies (the bias) and to the wide of the limits of agreement obtained will allow to select the best observer between the technician and the pulmonologist.

After the validation of the 3D-IC measurement against spirometry (difference > 10%), and after having confirmed that this analysis can be performed in routine by a pulmonary function technician, the next step will be to validate that the decrease of abdominal contribution of 3D-IC is an non-invasive index of diaphragmatic dysfunction. Accordingly, a linear regression analysis will be used in this study between the abdominal contribution to 3D-IC and the other parameters issued from exams prescribed by the clinician to confirm and evaluate diaphragmatic dysfunction. These other parameters are usually the fall of CV in supine position and/or a decrease of transdiaphragmatic pressure (Pdi) measurement by estimating the difference between oesophageal pressure (Peso) (intrathoracic pressure) and gastric pressure (Pga) (intra-abdominal pressure), [Pdi=Pga-Peso]. Pdi can be obtained during maximal voluntary efforts (the most frequent being the sniff test (Sniff Pdi)) or by using non-volitional test such as magnetic stimulation of the phrenic nerves (Twitch Pdi).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 90 years of age;
* Patients addressed for suspicion of diaphragmatic dysfunction, and able to maintain 5 sec of apnea in supine position.

Exclusion Criteria:

* Decubitus impossible;
* Apnea of 5 seconds impossible;
* Pregnant or Breastfeeding;
* Patient under juridic protection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients addressed to the respiratory function laboratory for suspicion of diaphragmatic dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Inspiratory capacity using a 3D technique | at baseline
  Thoraco-abdominal volume difference between the two respiratory positions will be calculated to obtain a difference in respiratory volume between these two positions.

SECONDARY OUTCOMES:
Abdominal contribution to inspiratory capacity | at baseline
  Abdominal contribution to trunck volume change

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric LOFASO, MD, PhD, Study Director — Physiological/Respiratory functional exploration Department, Raymond Poincaré Hospital, APHP; Caroline HELIE, Principal Investigator — Physiological/Respiratory functional exploration Department, Raymond Poincaré Hospital, APHP
Locations (1):
- Physiological/Respiratory functional exploration Department, Raymond Poincaré Hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No